## Generalized Anxiety Disorder Clinical Trials: An Analysis Regarding Engagement Trends and Participation of Generalized Anxiety Disorder Patients Involved in Clinical Trials

An Informed Consent Form For <u>Power Clinical Trial's</u>
Observational Study Involving Patients in Generalized Anxiety
Disorder Clinical Trials

Date: February 2, 2024

Introduction to Informed Consent Procedure: A Comprehensive Overview

This brief description seeks to offer an overview of our observational clinical investigation, emphasizing the protocols, potential risks, and advantages for participants. While your consent is required, your participation is fully optional, allowing you to withdraw without repercussions.

Our study seeks to understand the factors that influence generalized anxiety disorder patients' decisions to participate, persist, or discontinue in clinical trials. The primary processes include completing surveys and making follow-up calls, which are rigorously planned to reduce any hazards to participants.

Though immediate medical benefits may not be obvious in this observational study, the collected data will be critical in determining measures to increase clinical trial participation rates, ultimately helping patients suffering from generalized anxiety disorder.

The study's findings will provide critical insights into the factors influencing clinical trial participation rates. Our goal is to improve recruiting tactics and increase patient involvement in trials, resulting in better treatment options and results for people with

generalized anxiety disorder. It is crucial to remember that participation is entirely optional.

Before making a choice, make sure to properly understand the consent form and get clarity on any issues. It is recommended that you consult with your family, friends, advisers, and healthcare specialists to make an educated decision.

Factors Influencing Engagement in Clinical Studies on Generalized Anxiety Disorder

Clinical trials are pivotal for advancing generalized anxiety disorder treatments, yet questions persist about the varied representation of participants. This inquiry scrutinizes the determinants impacting patient decisions regarding their initiation, withdrawal, or re-involvement in generalized anxiety disorder clinical trials. Uncovering these determinants is crucial for refining the relevance and efficacy of future research initiatives.

To foster a comprehensive understanding, our emphasis is on recruiting a diverse demographic. We aim to unravel how variables such as age, race, income, and education mold decisions about participation. The collected data aspires to devise more effective strategies for engaging underrepresented groups in forthcoming clinical trials.

Participation in this study is entirely voluntary, granting individuals the liberty to withdraw without facing consequences. The study's procedures, including questionnaire completion and follow-up calls, entail minimal risks. Prospective participants are strongly encouraged to thoroughly scrutinize the consent form and seek clarification for any inquiries.

Ultimately, this trial seeks to deepen our comprehension of the determinants influencing participation in generalized anxiety disorder clinical trials. Improving participation rates could hasten the development of innovative treatments for this challenging ailment.

Exploring the Engagement Patterns of Individuals with Generalized Anxiety Disorder in Clinical Trials

Our observational clinical investigation aims to unravel the nuanced factors influencing the decision-making process of individuals with generalized anxiety disorder regarding their involvement in clinical trials, whether it be enrollment, withdrawal, or completion. Actively seeking volunteers from ongoing or concluded interventional studies, we leverage electronic medical records to identify potential participants.

Upon expressing interest, participants receive a comprehensive consent form outlining the study's objectives and participant rights. Biweekly questionnaires, delving into demographics, medical history, and factors affecting trial participation, serve as a primary data collection method. Additionally, we aspire to conduct thorough quarterly phone or video interviews to gain valuable insights from participants.

The statistical analysis of the gathered data endeavors to unveil the multifaceted factors influencing patient engagement in clinical trials. Our research findings will be disseminated through conferences and scholarly papers, benefiting all stakeholders involved in clinical trials.

These discoveries will contribute to shaping the future design of clinical trials for individuals with generalized anxiety disorder, alongside improving recruitment techniques and retention rates.

Participation in this study is entirely voluntary, allowing subjects the option to withdraw at any time without facing repercussions. The completion of surveys and follow-up interviews poses minimal risks, with our readily available research staff poised to promptly address any questions or concerns.

Evaluating Potential Hazards in Observational Research on Generalized Anxiety Disorder

Engaging in observational studies centered around generalized anxiety disorder does not involve participants in experimental treatments, yet it carries inherent risks. These risks encompass potential privacy breaches, emotional distress stemming from the study's subject matter, and possible adverse outcomes resulting from trial-related procedures.

Before committing to participation, it is imperative to thoroughly scrutinize and comprehend the informed consent form, addressing any concerns with the research team. The team is dedicated to furnishing comprehensive information regarding potential risks, the study's benefits, and the safety protocols in place to safeguard participants.

Investigating the Advantages of Engaging in Observational Trials for Generalized Anxiety Disorder

Participating in observational clinical trials focusing on generalized anxiety disorder provides patients with a chance to contribute to the progression of medical knowledge and potentially enhance future treatment alternatives. Despite the absence of experimental therapies, participants can avail themselves of comprehensive care throughout the study period.

Before deciding on trial participation, patients are urged to thoroughly assess potential benefits and risks, taking into account their circumstances and objectives. Seeking advice from healthcare providers and the research team becomes essential for making a well-informed decision.

Key Considerations Influencing Your Decision to End Participation

Acknowledging that your involvement in a clinical trial may terminate without your explicit consent is of significant importance. Researchers or sponsors may conclude the trial for various reasons, including study suspension, discontinuation of funding, or if it is deemed beneficial for your overall well-being.

Moreover, your participation might cease due to declining health, pregnancy, withdrawal after substantial updates, or non-compliance with study guidelines. Reflecting on these factors thoughtfully before committing to clinical trial participation is crucial.

An In-Depth Exploration of Various Trials Addressing Generalized Anxiety Disorder

Engaging in clinical studies related to generalized anxiety disorder is entirely voluntary, affording participants the option to withdraw without facing consequences.

Clinicaltrials.gov, overseen by the National Institutes of Health (NIH), stands as an extensive repository of active studies, providing a comprehensive overview of global research on generalized anxiety disorder. Users can customize their search based on their geographical location and specific medical concerns.

Moreover, Power's reference page offers an updated roster of presently ongoing generalized anxiety disorder clinical trials targeting actively seeking volunteers.

## Navigating the Landscape of Online Diversity in Clinical Trials

Numerous online platforms cater to individuals seeking profound insights into the diversity of clinical trials. Here are a couple of noteworthy articles that may capture your interest:

Mak, Winnie WS, Rita W. Law, Jennifer Alvidrez, and Eliseo J. Pérez-Stable. "Gender and ethnic diversity in NIMH-funded clinical trials: Review of a decade of published research." Administration and Policy in Mental Health and Mental Health Services Research 34 (2007): 497-503.

Joseph, Galen, and Daniel Dohan. "Diversity of participants in clinical trials in an academic medical center: the role of the 'Good Study Patient?'." Cancer 115, no. 3 (2009): 608-615.

These resources offer valuable insights into the challenges associated with achieving diversity in clinical trials and suggest potential strategies to foster inclusivity within research studies.

## Ensuring Data Privacy in Research Endeavors

Our foremost commitment is to safeguard the confidentiality of the data collected in the course of this research initiative. While achieving absolute confidentiality is not universally guaranteed, we have implemented robust measures to ensure its protection. It's crucial to acknowledge that legal obligations may, on occasion, necessitate the disclosure of personal information. Nevertheless, any research publications or presentations will prioritize your anonymity by abstaining from disclosing your name or any personally identifying information.

Entities such as accrediting bodies, government regulatory authorities (such as the FDA and OHRP), safety monitors, study sponsors, and authorized representatives may access your medical information for purposes related to research, quality assurance, and data analysis.

In exceptional cases, we may request an "Authorization Form" outlining the utilization and sharing of your information for this study. Prior to sharing your information or research samples with Power researchers, other university institutions, or external commercial entities for future research, explicit consent will be sought. Your confidential data will be handled securely and erased as appropriate.

Acknowledging Consent: Grasping the Stipulations

By endorsing this consent agreement, you acknowledge and accept the following terms:

- Thoroughly perusing and comprehending this informed consent form, with encouragement to explore alternative viewpoints before arriving at a decision.
- Ensuring satisfactory resolution of all your inquiries regarding the research project and its methodologies, equipping you with the necessary information for study participation.
- Deliberating on potential benefits, drawbacks, and alternatives associated with your involvement in the research.
- Receiving assurance that your voluntary participation in the research study will not impede your legal rights.
- Being assured of timely communication of any significant updates that might influence your decision to continue participating in the research study.

The receipt of this consent form offers you the opportunity to address any lingering inquiries.

| Participant's Signature | | |
|-------------------------|--------------------------|------|
| Name of Participant | Signature of Participant | Date |

| Researcher's Affirmation |
|---|
| In my role as the researcher, I assume the responsibility of addressing the patient's inquiries comprehensively, ensuring a thorough understanding of the study. Additionally, I reaffirm that the patient's participation is both voluntary and based on informed consent. |
| Signature of Researcher Who Received Consent |

Name of Investigator

Signature of Investigator Date